CLINICAL TRIAL: NCT07118683
Title: BRAZILIAN REGISTRY OF CHRONIC NON-COMMUNICABLE DISEASES IN PEOPLE LIVING WITH HIV/AIDS
Acronym: BRAVO
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Victor Augusto Hamamoto Sato, Principal Investigator, Hospital Alemão Oswaldo Cruz
Other Study IDs: CAAE: 81912924.9.1001.0070
Record Dates: First submitted 2025-07-06; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: AIDS (Acquired Immunodeficiency Syndrome); Cardiovascular and Cerebrovascular Diseases; Respiratory Comorbidities; Chronic Kidney Disease; Cancer
Keywords: Acquired Immunodeficiency Syndrome; Cardiovascular Diseases; Respiratory Tract Diseases; Renal Insufficiency, Chronic; Neoplasms; Treatment Adherence and Compliance; Quality of Life; Prevalence; Incidence; Brazil; Cross-sectional study; Prospective cohort
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cerebrovascular Disorders; Renal Insufficiency, Chronic; Neoplasms; Cardiovascular Diseases; Respiratory Tract Diseases; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BRAVO proposes the establishment of a comprehensive registry of chronic noncommunicable diseases (NCDs), providing crucial data for the formulation of effective health policies for people living with HIV/AIDS (PLWHA). The study will comprise a cross-sectional and longitudinal assessment: the cross-sectional study, will collect on the study allocation sociodemographic data, risk factors related to the main NCDs, physical examination data and samples for determination of biochemical and metabolic parameters; the longitudinal study, lasting 1 year and with the possibility of extension, will follow the participants to identify new diagnoses in the broad spectrum of NCDs. To this end, the study will include co-participating research centers from the 5 Brazilian geographic macro-regions.

DETAILED DESCRIPTION:
The BRAVO is a multicenter observational study. It includes a cross-sectional baseline assessment and a longitudinal cohort with annual follow-ups to evaluate cardiometabolic health, mental health, and quality of life among people living with HIV/AIDS (PLWHA).

BRAVO combines cross-sectional and prospective designs. Adults (≥18 years) with a confirmed HIV/AIDS diagnosis from across Brazil will be recruited in 2025, with follow-up starting in 2026. Participation requires informed consent. The cross-sectional phase captures data on risk factors, anthropometrics, and biological samples, while the longitudinal phase includes annual updates on clinical and mental health status, ART adherence, and quality of life (WHOQOL-BREF).

Data are collected using REDCap©, covering: i) Demographics and socioeconomic indicators; ii) Clinical and lab tests (cholesterol, HbA1c, triglycerides); iii) Physical measures (BMI, blood pressure, waist-hip ratio); iv) Respiratory (spirometry), renal, hepatic, and bone assessments (DXA); v) STIs, cancer risk, and CIMT (carotid ultrasound); vi) ART adherence (Morisky-Green), viral load, CD4/CD8 counts; vii) Mental health (depression, anxiety, substance use); and viii) Quality of life via WHOQOL-BREF.

Both validated and project-developed instruments will assess risk factors and outcomes. While validated tools improve reliability, the use of unvalidated questionnaires in certain domains (e.g., interpersonal violence) may introduce bias.

Regarding the sample size, the cross-sectional should include 79-310 participants (to detect diabetes prevalence); and the longitudinal should include 1,613-1,893 participants (to detect associations with risk factors), with a target of 2,100 participants considering dropouts.

Statistical Analysis Cross-sectional analysis uses standard tests (Chi-square, t-test, ANOVA, logistic regression) with methods for handling non-normal data and multivariable modeling.

Longitudinal data will be analyzed with paired tests (e.g., McNemar, paired t-test), GEE models, and ANCOVA. Missing data >5% will be imputed using machine learning (Orange software).

Subgroup analyses are planned for key populations (e.g., transgender, Black individuals, cisgender women).

Challenges No retention strategies are currently outlined, which could affect the study's internal validity due to participant attrition over time. Best practices like reminders and engagement initiatives are recommended.

Ethics The protocol has received approval from the Hospital Alemão Oswaldo Cruz ethics committee (CAAE: 7.003.613). Informed consent and participant confidentiality are ensured.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over;
* Any gender identity;
* Confirmed HIV or AIDS diagnosis;
* Signature of consent form

Exclusion Criteria:

* Indigenous population or those in prison in open or closed regimes;
* Patients hospitalized at the time of signing the Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV or Aids.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevelance of chronic non-communicable diseases and mental disorders | Baseline
  Prevalence of cardiovascular diseases, non-infectious respiratory diseases, chronic kidney disease and cancers, depression, dependence on alcohol and illicit substances, self-harm and physical violence.
Incidence of chronic non-communicable diseases and mental disorders | 1 year
  Cardiovascular diseases, non-infectious respiratory diseases, chronic kidney disease and cancers, and depression.

SECONDARY OUTCOMES:
Prevalence of metabolic and behavioral risk factors for chronic non-communicable diseases | Baseline
  History of hypertension, diabetes mellitus, dyslipidemia, smoking, physical activity, use of illicit drugs, alcoholism, dietary risk and continuous use medications, measurement of blood pressure, weight, height, abdominal and hip circumference, CD4, CD8, fasting blood glucose, HbA1C, total cholesterol and fractions, triglycerides, apolipoprotein A and B, serum and urinary creatinine, cystatin-C, urine 1, urinary albumin, serum and urinary phosphorus, urinary macroglobulin, urinary retinol-binding protein, AST, AST, Hepatitis A, B and C serologies, bone densitometry parameters, carotid ultrasound and spirometry.
Prevalence of participants with good adherence to antiretroviral therapy. | Baseline and 1 year after
  Adherence to antiretroviral therapy will be assessed using the 8-item Morisky-Green tool adapted for patients with HIV/AIDS.
  The instrument consists of eight dichotomous items. The questions were formulated to avoid a 'yes-saying' bias, so one point is assigned to each 'no' answer, except in item 5, which is reversed. At the end, patients are classified according to the score obtained as low adherers (score <6), medium adherers (score 6 to <8) and high adherers (score 8). The original authors also proposed a dichotomous cut-off of low (score <6) vs. high/medium adherence (score ≥6) to facilitate statistical analysis.
Profile of Quality of life of participants | Baseline and 1 year after
  Quality of life will be assessed by WHOQOL-BREF. The WHOQOL-BREF, a shortened version of the WHOQOL-100, is a 26-item questionnaire used to assess an individual's quality of life. It categorizes responses into four domains: Physical Health, Psychological Health, Social Relationships, and Environment. Each domain, along with the overall quality of life and general health questions, is scored on a 5-point Likert scale, which is then transformed to a 0-100 scale. A score of 100 represents the best possible quality of life within that domain.

OTHER OUTCOMES:
Incidence of adverse events potentially associated with antiretroviral therapy | Baseline and 1 year after
  Estimate adverse events potentially associated with antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Victor Sato, Principal Investigator — Hospital Alemão Oswaldo Cruz

IPD SHARING:
Plan to Share IPD: Undecided